CLINICAL TRIAL: NCT01133990
Title: An Open-Label, Multicenter, Randomized Phase Ib/II Study of FOLFIRI Alone Versus FOLFIRI Plus Bevacizumab Versus FOLFIRI Plus E7820 as Second-Line Therapy in Patients With Locally Advanced or Metastatic Colorectal Cancer
Brief Title: FOLFIRI Alone Versus FOLFIRI Plus Bevacizumab Versus FOLFIRI Plus E7820 as Second-Line Therapy in Patients With Locally Advanced or Metastatic Colorectal Cancer
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: The study was terminated early as the combination of E7820 and FOLFIRI was deemed to be not tolerable, hence no efficacy analysis was conducted.
Sponsor: Eisai Inc. (Industry)
Collaborators: Quintiles, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: E7820-701; 2009-016015-37 (EudraCT Number)
Record Dates: First submitted 2010-05-21; First posted 2010-05-31 (Estimated); Results first posted 2023-11-07 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2012-07

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — IFL protocol; Leucovorin; Fluorouracil; Irinotecan; N-(3-cyano-4-methyl-1H-indol-7-yl)-3-cyanobenzene-sulfonamide; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- FOLFIRI (Active Comparator): The FOLFIRI regimen consists of irinotecan at 180 mg/m2 (IV infusion) on Day 1 and Day 15 of each 28-day cycle, leucovorin at 200 mg/m2 (400 mg/m2 if using d,l-racemic mixture of leucovorin) by IV infusion on Days 1 and 15 of each cycle, and 5-FU at 400 mg/m2 as an IV bolus injection followed by a total of 2400 mg/m2 by CIV infusion over 46 hours over Days 1 and 2 via an ambulatory programmable pump (the use of an ambulatory pump is optional). The 5-FU IV bolus (400 mg/m2) and CIV infusion (2400 mg/m2) over 46 hours is repeated on Days 15 and 16 of each cycle.
  Interventions: Drug: FOLFIRI
- E7820 (Experimental): E7820 is administered orally in tablet form once daily, every day of each 28-day treatment cycle. For the Phase Ib portion, the doses will be 40 mg/day, 70 mg/day, and 100 mg/day, and for the Phase II portion, the dose will be the MTD recommended Phase IB dose in combination with FOLFIRI, as determined during the Phase Ib portion of the study.
  Interventions: Drug: FOLFIRI; Drug: E7820
- FOLFIRI plus Bevacizumab (Experimental): Bevacizumab at 5 mg/kg (IV infusion) on Days 1 and 15 of each 28-day treatment cycle
  Interventions: Drug: FOLFIRI; Drug: Bevacizumab

INTERVENTIONS:
Drug: FOLFIRI — FOLFIRI will be administered as IV infusion on Days 1 and 15 of each cycle, and 5-FU at 400 mg/m^2 as an IV bolus injection followed by a total of 2400 mg/m2 by CIV infusion over 46 hours over Days 1 and 2 via an ambulatory programmable pump. The 5-FU IV bolus (400 mg/m^2) and CIV infusion (2400 mg/m^2) over 46 hours is repeated on Days 15 and 16 of each cycle.
  Other Names: leucovorin calcium (calcium folinate), 5-fluorouracil, and irinotecan
Drug: E7820 — E7820 will be administered orally in tablet form once daily, every day of each 28-day treatment cycle.
  Arms: E7820
Drug: Bevacizumab — Bevacizumab will be administered at 5 mg/kg (IV infusion) on Days 1 and 15 of each 28-day treatment cycle.
  Other Names: Avastin
  Arms: FOLFIRI plus Bevacizumab

SUMMARY:
The purpose of the Phase Ib portion is to find out the highest dose of study drug that can safely be given when tested in a small group of subjects.

The purpose of the Phase II portion is to find out how safe the study drug is when taken at the highest dose in a larger group of subjects.

DETAILED DESCRIPTION:
The primary purpose for Phase 1b: to determine the maximum tolerated dose (MTD) of E7820 recommended for Phase 2 when administered in combination with the FOLFIRI regimen (irinotecan, leucovorin, and 5-fluorouracil [5-FU]) in participants with locally advanced or metastatic colorectal cancer (mCRC) who have failed first-line therapy. Phase 2: to evaluate the safety and tolerability of E7820 administered in combination with the FOLFIRI regimen, compared with FOLFIRI alone and FOLFIRI plus bevacizumab, in patients with locally advanced or mCRC who have failed first-line therapy.

ELIGIBILITY:
Inclusion Criteria:

Patients may be entered in the study only if they meet all of the following criteria:

1. Male or female patient greater than or equal to 18 years of age;
2. Histologically or cytologically confirmed nonresectable locally advanced or metastatic colorectal adenocarcinoma;
3. Patients must have failed a first-line chemotherapy regimen for nonresectable locally advanced or mCRC (first-line bevacizumab is allowed). Patients randomized to the Phase Ib portion can have up to 3 total prior regimens (including adjuvant therapy in addition to treatment for advanced disease);
4. At least 1 site of measurable disease by the Response Evaluation Criteria in Solid Tumors (RECIST version 1.1) criteria;
5. Life expectancy of > 3 months;
6. Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) 0 or 1;
7. Patients must have adequate renal function as evidenced by serum creatinine <2 mg/dL and creatinine clearance >50 mL/minute per the Cockcroft and Gault formula;
8. Patients must have adequate bone marrow function as evidenced by absolute neutrophil count (ANC) >1.5 x 109/L, platelets >100 x 109/L, hemoglobin >9.0 g/dL (a hemoglobin <9.0 g/dL at Screening is acceptable if it is corrected to >9 g/dL by growth factor or transfusion prior to first dose);
9. Patients must have adequate liver function as evidenced by bilirubin <1.5 times the upper limit of the normal range (ULN), and alkaline phosphatase, alanine aminotransferase (ALT), and aspartate aminotransferase (AST) <3 X ULN (in the case of liver metastases, <5 X ULN). If there are bone metastases, liver-specific alkaline phosphatase may be separated from the total and used to assess liver function instead of total alkaline phosphatase;
10. Blood pressure must be well-controlled (<140/90 mmHg at screening) with or without antihypertensive medication. Patients must have no history of hypertensive crisis or hypertensive encephalopathy;
11. Male or female patients of child-producing potential must agree to use double barrier contraception, oral contraceptives, or avoidance of pregnancy measures during the study and for 90 days after the last day of treatment;
12. Females of childbearing potential must have a negative serum pregnancy test;
13. Females may not be breastfeeding; and
14. Ability to understand and willingness to sign a written consent.

Exclusion Criteria:

Patients will not be entered in the study for any of the following reasons:

1. Received chemotherapy, targeted therapy, radiotherapy, surgery, immunotherapy, or treatment in another clinical study within the 30 days prior to commencing study treatment or have not recovered from side effects of all treatment-related toxicities to Grade <1, except for peripheral neuropathy (Grade 1 and Grade 2 are permitted) and alopecia;
2. Previously received irinotecan or irinotecan derivatives;
3. Previously received anti-alpha 2 integrin therapy;
4. History of other malignancies except: (1) adequately treated basal or squamous cell carcinoma of the skin; (2) curatively treated, a) in situ carcinoma of the uterine cervix, b) prostate cancer, or c) superficial bladder cancer; or (3) other curatively treated solid tumor with no evidence of disease for >5 years;
5. Presence of brain metastases, unless the patient has received adequate treatment at least 4 weeks prior to randomization, and is stable, asymptomatic, and off steroids for at least 4 weeks prior to randomization;
6. Are currently receiving any other anticancer treatment;
7. Palliative radiotherapy is not permitted throughout the study period;
8. Serious non-healing wound, ulcer, or active bone fracture;
9. Major surgical procedure, open biopsy or significant traumatic injury within 28 days prior to Day 1, or anticipation of need for a major surgical procedure during the course of the study;
10. Refractory nausea and vomiting, malabsorption, significant bowel resection, or any other medical condition that would preclude adequate absorption or result in the inability to take oral medication;
11. Significant cardiovascular impairment (history of congestive heart failure New York Heart Association [NYHA] Grade >2, unstable angina or myocardial infarction within the past 6 months, or serious cardiac arrhythmia);
12. Active hemoptysis (defined as bright red blood of
13. Current or recent use (within 7 days) of full-dose warfarin (except low-dose warfarin as required to maintain patency of preexisting, permanent indwelling IV catheters). For subjects receiving warfarin, International Normalization Ratio (INR) should be <1.5. Patients may have prophylactic use of low molecular weight heparin, however therapeutic use of heparin or low molecular weight heparin is not acceptable;
14. History of bleeding diathesis or coagulopathy;
15. Any history of cerebral vascular accident, transient ischemic attack or ≥ Grade 2 peripheral vascular disease, unless they have had no evidence of active disease for at least 6 months prior to randomization;
16. Abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within 6 months prior to Day 1, unless affected area has been removed surgically;
17. Patients with organ allografts requiring immunosuppression;
18. Known positive human immunodeficiency virus (HIV), known hepatitis B surface antigen, or active hepatitis C positive;
19. Patients with a history of allergic reactions attributed to compounds of similar chemical or biologic composition to bevacizumab, irinotecan, 5-FU, or leucovorin;
20. Hypersensitivity to sulfonamide derivatives; or
21. Have any medical condition that would interfere with the conduct of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2010-03-04 (Actual); Primary Completion 2011-02-18 (Actual); Study Completion 2011-02-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Harish Dave, Study Director — Quintiles, Inc.
Locations (34):
- United States (6):
  - Rocky Mountain Cancer Center - Midtown, Denver, Colorado
  - Summit Medical Group, Berkeley Heights, New Jersey
  - Hematology Oncology Associates SJ P.A., Mount Holly, New Jersey
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Northwest Medical Specialties, PLLC, Tacoma, Washington
- Australia (9):
  - North Coast Cancer Institute, Coffs Harbour, New South Wales
  - Sydney Haematology & Oncology Clinic, Hornsby, New South Wales
  - Calvary Mater Newcastle, Waratah, New South Wales
  - Royal Brisbane and Women's Hospital, Herston, Queensland
  - Royal Hobart Hospital, Hobart, South Australia
  - Queen Elizabeth Hospital, Woodville South, South Australia
  - Box Hill Hospital, Box Hill, Victoria
  - The Austin Hospital, Epping, Victoria
  - Newcastle Private Hospital, Merewether
- India (10):
  - Jawaharlal Nehru Cancer Hospital and Research Centre, Bhopal, Madhya Pradesh
  - Searoc Cancer Hosptial, Jaipur, Rajasthan
  - Gujarat Cancer & Research Institute, Ahmedabad
  - Kidwai Institute of Oncology, Bangalore
  - M. S. Ramaiah Memorial Hospital, Bangalore
  - Subodh Mitra Cancer Hospital and Research centre, Kolkata
  - Shatabdi Hospital, Nashik
  - Deenanath Mangeshkar Hospital and Research Center, Pune
  - Noble Hospital, Pune
  - Christian Medical College, Vellore
- Russia (4):
  - CCH #2 n.a. N. A. Semashko of LLC "Russian Railways", Moscow
  - City Mariinskaya Hospital, Saint Petersburg
  - Scientific Research Oncology Institute named after N.N. Petr, Saint Petersburg
  - Yaroslav Regional Clinical Oncology Hospital, Yaroslav
- Ukraine (5):
  - Mun. Multifield Clin.Hosp.#4,Dept. of Chemotherapy, DSMU, Dnipropetrovsk
  - Donetsk Regional Anticancer Centre, Donetsk
  - City Clinical Hospital #2, Kharkiv
  - The St.Inst. "S.P.Grigoriev Med. Rad.Inst. of AMS of Ukr.", Kharkiv
  - Uzhgorod Centr.City Cl.Hosp.,City Onc.Center, UNMU,Fac.of PG, Uzhhorod

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 4 investigative sites in Australia and the United States from 04 March 2010 to 18 February 2011.
Pre-assignment Details: A total of 5 participants were enrolled and treated in Phase 1b part of the study and only safety was analyzed for all participants in this study. The planned dose escalation of E7820 at 70 milligram per day (mg/day), 100 mg/day and Phase 2 part were not conducted as the study was terminated early without determination of the Maximum Tolerated Dose (MTD) as the combination of E7820 plus FOLFIRI (irinotecan, leucovorin, and 5-fluorouracil [5-FU]) was deemed to be not tolerable.
Groups:
- Phase 1b: E7820 40 mg/Day + FOLFIRI: Participants received E7820 40 mg/day tablets orally, in combination with a FOLFIRI regimen on Days 1 to 2 and 15 to 16 of each 28-day treatment cycle. FOLFIRI regimen consisted of; Irinotecan 180 milligram per square meter (mg/m^2), Leucovorin 200 mg/m^2 administered by intravenous (IV) infusion on Days 1 and 15 of each 28-day treatment cycle, and 400 mg/m^2 5-fluorouracil (5-FU) administered as an IV bolus injection followed by a total of 2400 mg/m^2 5-FU administered by continuous IV (CIV) infusion over 46 hours on Days 1 to 2, then repeated on Days 15 to 16 of each 28-day treatment cycle. Participants continued to receive study treatment unless there was occurrence of progressive disease (PD), unacceptable toxicity, withdrawal of consent, withdrawal by the investigator, lost to follow-up, or death, whichever occurred first.
- Phase 1b: E7820 70 mg/Day + FOLFIRI; Phase 2: E7820 (RP2D) + FOLFIRI: Participants were planned to receive E7820 70 mg/day tablets orally, in combination with a FOLFIRI regimen on Days 1 to 2 and 15 to 16 of each 28-day treatment cycle. FOLFIRI regimen consisted of; Irinotecan 180 mg/m^2, Leucovorin 200 mg/m^2 administered by IV infusion on Days 1 and 15 of each 28-day treatment cycle, and 400 mg/m^2 5-FU administered as an IV bolus injection followed by a total of 2400 mg/m^2 5-FU administered by CIV infusion over 46 hours on Days 1 to 2, then repeated on Days 15 to 16 of each 28-day treatment cycle. Participants were planned to receive study treatment unless there was occurrence of PD, unacceptable toxicity, withdrawal of consent, withdrawal by the investigator, lost to follow-up, or death, whichever occurred first. No participants were enrolled in this arm. The study did not progress beyond Phase 1b (E7820 40 mg/day).
- Phase 1b: E7820 100 mg/Day + FOLFIRI: Participants were planned to receive E7820 100 mg/day tablets orally, in combination with a FOLFIRI regimen on Days 1 to 2 and 15 to 16 of each 28-day treatment cycle. FOLFIRI regimen consisted of; Irinotecan 180 mg/m^2, Leucovorin 200 mg/m^2 administered by IV infusion on Days 1 and 15 of each 28-day treatment cycle, and 400 mg/m^2 5-FU administered as an IV bolus injection followed by a total of 2400 mg/m^2 5-FU administered by CIV infusion over 46 hours on Days 1 to 2, then repeated on Days 15 to 16 of each 28-day treatment cycle. Participants were planned to receive study treatment unless there was occurrence of PD, unacceptable toxicity, withdrawal of consent, withdrawal by the investigator, lost to follow-up, or death, whichever occurred first. No participants were enrolled in this arm. The study did not progress beyond Phase 1b (E7820 40 mg/day).
- Phase 2: FOLFIRI: Participants were planned to receive FOLFIRI regimen consisted of; Irinotecan 180 mg/m^2, Leucovorin 200 mg/m^2 administered by IV infusion on Days 1 and 15 of each 28-day treatment cycle, and 400 mg/m^2 5-FU administered as an IV bolus injection followed by a total of 2400 mg/m^2 5-FU administered by CIV infusion over 46 hours on Days 1 to 2, then repeated on Days 15 to 16 of each 28-day treatment cycle. Participants were planned to receive study treatment unless there was occurrence of PD, unacceptable toxicity, withdrawal of consent, withdrawal by the investigator, lost to follow-up, or death, whichever occurred first. No participants were enrolled in this arm. The study did not progress beyond Phase 1b (E7820 40 mg/day).
- Phase 2: FOLFIRI + Bevacizumab: Participants were planned to receive FOLFIRI regimen consisted of; Irinotecan 180 mg/m^2, Leucovorin 200 mg/m^2 administered by IV infusion on Days 1 and 15 of each 28-day treatment cycle, and 400 mg/m^2 5-FU administered as an IV bolus injection followed by a total of 2400 mg/m^2 5-FU administered by CIV infusion over 46 hours on Days 1 to 2, then repeated on Days 15 to 16 of each 28-day treatment cycle followed by Bevacizumab 5 mg/kg, IV infusion on Days 1 and 15 of each 28-day treatment cycle. Participants were planned to receive study treatment unless there was occurrence of PD, unacceptable toxicity, withdrawal of consent, withdrawal by the investigator, lost to follow-up, or death, whichever occurred first. No participants were enrolled in this arm. The study did not progress beyond Phase 1b (E7820 40 mg/day).
Period: Phase 1b (Dose Escalation Phase)
Arm/Group | Phase 1b: E7820 40 mg/Day + FOLFIRI | Phase 1b: E7820 70 mg/Day + FOLFIRI | Phase 1b: E7820 100 mg/Day + FOLFIRI | Phase 2: FOLFIRI | Phase 2: FOLFIRI + Bevacizumab | Phase 2: E7820 (RP2D) + FOLFIRI
Started | 5 | 0 | 0 | 0 | 0 | 0
Completed | 1 | 0 | 0 | 0 | 0 | 0
Not Completed | 4 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Progression of disease | 1 | 0 | 0 | 0 | 0 | 0
Period: Phase 2 (Dose-confirmation Phase)
Arm/Group | Phase 1b: E7820 40 mg/Day + FOLFIRI | Phase 1b: E7820 70 mg/Day + FOLFIRI | Phase 1b: E7820 100 mg/Day + FOLFIRI | Phase 2: FOLFIRI | Phase 2: FOLFIRI + Bevacizumab | Phase 2: E7820 (RP2D) + FOLFIRI
Started (The study was terminated after phase 1b (E7820 40 mg/day). Hence, no participants were enrolled in Phase 2.) | 0 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety population included all participants who received at least one dose of study drug and who had safety assessment post the first dose.
Groups:
- Phase 1b: E7820 40 mg/Day + FOLFIRI: Participants received E7820 40 mg/day tablets orally, in combination with a FOLFIRI regimen on Days 1 to 2 and 15 to 16 of each 28-day treatment cycle. FOLFIRI regimen consisted of; Irinotecan 180 mg/m^2, Leucovorin 200 mg/m^2 administered by IV infusion on Days 1 and 15 of each 28-day treatment cycle, and 400 mg/m^2 5 -FU administered as an IV bolus injection followed by a total of 2400 mg/m^2 5-FU administered by CIV infusion over 46 hours on Days 1 to 2, then repeated on Days 15 to 16 of each 28-day treatment cycle. Participants continued to receive study treatment unless there was occurrence of PD, unacceptable toxicity, withdrawal of consent, withdrawal by the investigator, lost to follow-up, or death, whichever occurred first.
Arm/Group | Phase 1b: E7820 40 mg/Day + FOLFIRI
Number analyzed (Participants) | 5
Age, Customized [Count of Participants; unit: Participants]
  43 - 83 years | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 4
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 5
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Phase 1b: Number of Participants With Dose-limiting Toxicities (DLTs)
Description: Dose-limiting toxicities were defined as clinically significant adverse events (AEs) occurring less than or equal to (<=) 28 days after commencing study treatment and considered by the investigator to be possibly or probably related to study treatment. Toxicity was evaluated according to National Cancer Institute Common Terminology Criteria for Adverse Events version 4.0 (NCI CTCAE v.4.0).
Time Frame: Cycle 1 (each cycle length=28 days)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1b: E7820 40 mg/Day + FOLFIRI
Number analyzed (Participants) | 5
Participants | 2

2. Primary Outcome: Phase 1b: Number of Participants With Any Treatment-emergent Adverse Events (TEAEs)
Description: Adverse Events were defined as TEAEs if they started on or after the date and time of administration of the first dose of study drug during the study. An AE was defined as any untoward medical occurrence in a participant administered a pharmaceutical product, and which did not necessarily have a causal relationship with this treatment. Any change in hematology, clinical chemistry, urine values and regular measurement of vital signs which were deemed clinically significant by the investigator were recorded as TEAE.
Time Frame: From date of first dose up to 30 days after last dose of study treatment (up to 11.5 months)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1b: E7820 40 mg/Day + FOLFIRI
Number analyzed (Participants) | 5
Participants | 5

3. Primary Outcome: Phase 1b: Number of Participants With Eastern Cooperative Oncology Group Performance Status (ECOG-PS)
Description: ECOG-PS measured participant's performance status on 5 point scale: 0=Fully active/able to carry on all pre-disease activities without restriction; 1=restricted in physically strenuous activity, ambulatory/able to carry out light or sedentary work; 2=ambulatory (greater than[ >] 50 percent [%] of waking hours), capable of all self care, unable to carry out any work activities; 3=capable of only limited self care, confined to bed/chair >50% of waking hours; 4=completely disabled, cannot carry on any self care, totally confined to bed/chair; 5=dead.
Time Frame: From date of first dose up to 30 days after last dose of study treatment (up to 11.5 months)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1b: E7820 40 mg/Day + FOLFIRI
Number analyzed (Participants) | 5
Participants
  Participants With ECOG-PS Grade 1 | 1
  Participants With ECOG-PS Grade 2 | 2
  Participants With ECOG-PS Grade 3 | 2
  Participants With ECOG-PS Grade 4 | 0
  Participants With ECOG-PS Grade 5 | 0

4. Primary Outcome: Phase 1b: Number of Participants With Clinically Significant Changes in Physical Examinations
Description: Physical examination included examination of the head, eyes, ears, nose, throat, neck, heart, chest, lungs, abdomen, extremities, skin, lymph nodes, and neurological status.
Time Frame: From date of first dose up to 30 days after last dose of study treatment (up to 11.5 months)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1b: E7820 40 mg/Day + FOLFIRI
Number analyzed (Participants) | 5
Participants | 2

5. Primary Outcome: Phase 1b: Number of Participants With Clinically Significant Change From Baseline in Electrocardiograms (ECGs) Parameter
Description: ECG was to be a complete standardized 12-lead recording. The ECGs were reviewed by the investigator or designee prior to study drug administration as part of the participant's standard of care.
Time Frame: From date of first dose up to 30 days after last dose of study treatment (up to 11.5 months)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1b: E7820 40 mg/Day + FOLFIRI
Number analyzed (Participants) | 5
Participants | 1

6. Secondary Outcome: Phase 2: Progression-Free Survival (PFS)
Description: PFS was defined as the time from the date of randomization of a participant to the date of first documentation of PD or death (whichever occurred first) based on investigator assessments according to Response Evaluation Criteria in Solid Tumors (RECIST) version (v) 1.1. PD was defined as at least a 20% increase or 5 millimeter (mm) increase in the sum of diameters of target lesions (taking as reference the smallest sum on study) recorded since the treatment started or the appearance of 1 or more new lesions.
Time Frame: From the date of randomization to date of PD or death (whichever occurred first), up to 11 months
Population: The study was terminated before the initiation of Phase 2, so the data for this outcome measure was not collected and analyzed.
Arm/Group | Phase 2: FOLFIRI | Phase 2: FOLFIRI + Bevacizumab | Phase 2: E7820 (RP2D) + FOLFIRI
Number analyzed (Participants) | 0 | 0 | 0

7. Secondary Outcome: Phase 2: Time to Progression (TTP)
Description: TTP was defined as time from the date of randomization of a participant until the date of first documented progression of such participant's disease based on investigator assessments according to RECIST v.1.1. PD was defined as at least a 20% increase or 5 mm increase in the sum of diameters of target lesions (taking as reference the smallest sum on study) recorded since the treatment started or the appearance of 1 or more new lesions.
Time Frame: From date randomization to date of PD or death, up to 11 months
Population: as for outcome 6
Arm/Group | Phase 2: FOLFIRI | Phase 2: FOLFIRI + Bevacizumab | Phase 2: E7820 (RP2D) + FOLFIRI
Number analyzed (Participants) | 0 | 0 | 0

8. Secondary Outcome: Phase 2: Objective Response Rate (ORR)
Description: ORR was defined as percentage of participants in the study whose best overall response was either CR or PR based on investigator assessments according to RECIST v1.1. A confirmatory scan was required after no less than 4 weeks and no later than 8 weeks, starting on the date that the response was first recorded. CR was defined as the disappearance of all target and non-target lesions (non-lymph nodes). All pathological lymph nodes (whether target or non-target) must have a reduction in their short axis to less than (<)10 mm. PR was defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: From date of treatment start to until date of first PD or death (whichever occurred first), up to 11 months
Population: as for outcome 6
Arm/Group | Phase 2: FOLFIRI | Phase 2: FOLFIRI + Bevacizumab | Phase 2: E7820 (RP2D) + FOLFIRI
Number analyzed (Participants) | 0 | 0 | 0

9. Secondary Outcome: Phase 2: Overall Survival (OS)
Description: OS was defined as time from the date of randomization of a participant until the date of death of such participant, regardless of the actual cause of the participant's death.
Time Frame: From date of randomization to date of PD or death, up to 11 months
Population: as for outcome 6
Arm/Group | Phase 2: FOLFIRI | Phase 2: FOLFIRI + Bevacizumab | Phase 2: E7820 (RP2D) + FOLFIRI
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Phase 1b: From date of first dose up to 30 days after last dose of study treatment (up to 11.5 months)
Arm/Group | Phase 1b: E7820 40 mg/Day + FOLFIRI
All-Cause Mortality (participants affected / at risk) | 2/5
Serious Adverse Events (participants affected / at risk) | 2/5
Other Adverse Events (participants affected / at risk) | 5/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1b: E7820 40 mg/Day + FOLFIRI (N=5)
Sepsis (Infections and infestations) | 1
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1
Septic shock (Infections and infestations) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1b: E7820 40 mg/Day + FOLFIRI (N=5)
Fatigue (General disorders) | 3
Diarrhoea (Gastrointestinal disorders) | 2
Mucosal inflammation (General disorders) | 2
Neutropenia (Blood and lymphatic system disorders) | 2
Weight decreased (Investigations) | 2
Abdominal discomfort (Gastrointestinal disorders) | 1
Acute myocardial infarction (Cardiac disorders) | 1
Adverse drug reaction (General disorders) | 1
Alopecia (Skin and subcutaneous tissue disorders) | 1
Amnesia (Nervous system disorders) | 1
Anaemia (Blood and lymphatic system disorders) | 1
Ascites (Gastrointestinal disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Blister (Skin and subcutaneous tissue disorders) | 1
Chest pain (General disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Dizziness (Nervous system disorders) | 1
Dysgeusia (Nervous system disorders) | 1
Dyspepsia (Gastrointestinal disorders) | 1
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Dysuria (Renal and urinary disorders) | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Gastritis (Gastrointestinal disorders) | 1
Haematochezia (Gastrointestinal disorders) | 1
Leukopenia (Blood and lymphatic system disorders) | 1
Mouth ulceration (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Oedema (General disorders) | 1
Oedema peripheral (General disorders) | 1
Oesophagitis (Gastrointestinal disorders) | 1
Oral candidiasis (Infections and infestations) | 1
Orthostatic hypotension (Vascular disorders) | 1
Palpitations (Cardiac disorders) | 1
Pyrexia (General disorders) | 1
Stomatitis (Gastrointestinal disorders) | 1
Swelling face (Skin and subcutaneous tissue disorders) | 1
Syncope (Nervous system disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Venous occlusion (Vascular disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Vulvovaginal candidiasis (Infections and infestations) | 1

LIMITATIONS AND CAVEATS:
The study was terminated early as the combination of E7820 and FOLFIRI was deemed to be not tolerable, hence no efficacy analysis was conducted.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other